CLINICAL TRIAL: NCT04645342
Title: Wire Instrumentation Using Radiofrequency Energy to Impact Transseptal Efficiency
Acronym: WIRE-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Baylis Medical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-30738
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Results first posted 2023-03-10 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Baylis Versacross RF wire (Experimental): Device: Baylis Versacross radiofrequency wire
  Interventions: Device: Baylis Versacross RF wire
- Baylis RF Needle (Active Comparator): Device: conventional Baylis radiofrequency needle
  Interventions: Device: Baylis RF needle

INTERVENTIONS:
Device: Baylis Versacross RF wire — Baylis Versacross radiofrequency wire is used for transseptal puncture during cardiac ablation procedure.
  Arms: Baylis Versacross RF wire
Device: Baylis RF needle — Baylis radiofrequency needle is used for transseptal puncture during cardiac ablation procedure.
  Arms: Baylis RF Needle

SUMMARY:
This is a randomized controlled trial examining whether Baylis's Versacross RF wire versus the conventional Baylis RF needle is better at puncturing through a thin wall in the heart (called "transseptal puncture") as measured by time to successful transseptal puncture, during cardiac ablation procedures.

DETAILED DESCRIPTION:
The transseptal puncture is one of the most commonly performed procedures in the cardiac electrophysiology and interventional cardiology laboratories. Indeed, every atrial fibrillation ablation, now the predominant electrophysiology procedure performed throughout the world, routinely involves two different transseptal puncture procedures. The investigators previously performed a randomized, comparative effectiveness trial demonstrating the superiority (in both efficacy and safety) of a radiofrequency (RF) transseptal needle versus the conventional sharp-tipped mechanical needle. More recently, an alternative approach to transseptal puncture has been FDA approved and is already utilized as part of standard of care in these procedures. With this new approach, a J-shaped wire that can transmit RF energy is advanced inside the transeptal sheath rather than the more stiff RF or conventional needle. As advancing a wire is usually a step employed in any transseptal procedure (then usually requiring removal of that wire and then placement of the needle), this new approach saves a step. In addition once the wire has been advanced across the intra-atrial septum into the left atrium, the wire can be used to avoid potentially severe complications; specifically, after a transseptal needle is advanced across the left atrium, advancing the sheath over the needle can result in a sudden jump of all the equipment, risking perforation of the far left atrial wall. With the wire approach, the wire can be safely advanced into a pulmonary vein so that even if the sheath and dilator jump suddenly across the septum, they will be guided along the wire and thereby avoid perforation. The investigators will be studying patients undergoing a catheter ablation procedure at University of California, San Francisco.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patients undergoing endocardial left atrial catheter ablation procedures using radiofrequency ablation catheters for atrial fibrillation or atrial flutter ablation procedures at UCSF
* Willing and able to provide written informed consent in English
* Willing and able to comply with scheduled remote follow-up visits through 1 Year post-operative

Exclusion Criteria:

* Presence of a patent foramen ovale closure device or atrial septal defect closure device
* Cryoballoon ablation
* IVC filter
* Deemed not suitable by study personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Marcus, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 11/30/2020 to 2/2/2022, 75 participants were enrolled and randomized in the study.
Pre-assignment Details: 261 patients were assessed for eligibility; 61 declined to participate, 118 met exclusion criteria, 7 did not enroll for other reasons.
Period: Overall Study
Arm/Group | Baylis RF Needle | Baylis Versacross RF Wire
Started | 36 | 39
Completed | 36 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Baylis RF Needle: Device: conventional Baylis radiofrequency needle
  Baylis RF needle: Baylis radiofrequency (RF) needle is used for transseptal puncture during cardiac ablation procedure.
- Baylis Versacross RF Wire: Device: Baylis Versacross radiofrequency wire
  Baylis Versacross RF wire: Baylis Versacross radiofrequency (RF) wire is used for transseptal puncture during cardiac ablation procedure.
- Total: Total of all reporting groups
Arm/Group | Baylis RF Needle | Baylis Versacross RF Wire | Total
Number analyzed (Participants) | 36 | 39 | 75
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [57 to 69] | 61 [55 to 70] | 63 [55 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 28 | 29 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26 | 28 | 54
  Black | 1 | 2 | 3
  Asian | 5 | 5 | 10
  Other | 4 | 4 | 8
Height [Mean (Standard Deviation); unit: cm] | 177 (8) | 176 (9) | 176 (14)
Weight [Median (Inter-Quartile Range); unit: kg] | 86 [78 to 105] | 94 [75 to 113] | 91 [77 to 108]
Prior transseptal procedure [Count of Participants; unit: Participants] | 7 | 9 | 16
Paroxysmal atrial fibrillation/flutter [Count of Participants; unit: Participants] | 18 | 16 | 34
CHA2DS2VASC score [Median (Inter-Quartile Range); unit: scores on a scale (0-9)] — The acronym CHA2DS2-VASc stands for congestive heart failure, hypertension, age ≥75 (doubled), diabetes, stroke (doubled), vascular disease, age 65 to 74 and sex category (female). Two points are awarded for stroke, TIA or thromboembolism in the medical history and for age over 75. One point is assigned for age 65 to 75, Hypertension, diabetes mellitus, heart failure or ejection fraction <40%, vascular disease (prior myocardial infarction, peripheral artery disease, aortic plaque), and female sex. Score 0 - low risk, score 1 - medium risk, score ≥2 - high risk. Scores can range from 0-9.
  scores on a scale (0-9) | 3 [2 to 4] | 3 [2 to 4] | 3 [2 to 4]
Transvenous pacemaker or defibrillator [Count of Participants; unit: Participants] | 3 | 4 | 7
Left atrial size by transthoracic echocardiogram (TTE) [Count of Participants; unit: Participants]
  Normal | 12 | 16 | 28
  Mild to moderately enlarged | 18 | 16 | 34
  Severely enlarged | 6 | 7 | 13
Rhythm at time of transseptal [Count of Participants; unit: Participants]
  Sinus or atrial paced | 21 | 21 | 42
  Atrial fibrillation or atrial flutter | 15 | 18 | 33

OUTCOME MEASURES:

1. Primary Outcome: Time to Achieve First Transseptal Puncture
Description: First transseptal time was recorded for each participant, starting with insertion of the long guidewire into the femoral short sheath (J wire for RF needle group, VersaCross wire for RF wire group) and stopping once the transseptal sheath was positioned in the LA and the dilator and guidewire were fully removed from the long sheath. Median time in minutes to completion of the first transseptal puncture during the cardiac ablation procedure between the RF needle and RF Wire group was compared as the outcome.
Time Frame: 0-30 minutes (from insertion of guidewire to removal of guidewire of first transseptal)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Baylis RF Needle | Baylis Versacross RF Wire
Number analyzed (Participants) | 36 | 39
minutes | 9.2 [5.7 to 11.2] | 6.9 [5.2 to 8.4]

2. Secondary Outcome: Time to Achieve Second Transseptal Puncture
Description: Second transseptal time was recorded for each participant, starting with insertion of the long guidewire into the femoral short sheath (J wire for RF needle group, VersaCross wire for RF wire group) and stopping once the transseptal sheath was positioned in the LA and the dilator and guidewire were fully removed from the long sheath. The median time in minutes to completion of the second transseptal puncture during the cardiac ablation procedure between the RF needle and RF Wire group was compared as a secondary outcome. Participants that did not undergo 2 transseptal punctures were not included in this analysis.
Time Frame: 0-30 minutes (from insertion of guidewire to removal of guidewire of second transseptal)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Baylis RF Needle | Baylis Versacross RF Wire
Number analyzed (Participants) | 30 | 35
minutes | 8.4 [5.5 to 13.4] | 6.0 [4.9 to 7.8]

3. Secondary Outcome: Combined Transseptal Time
Description: Combined transseptal time was calculated for each participant by summing up participants' first and second transseptal times. The median combined transseptal time in minutes between the RF needle and RF Wire group was compared as a secondary outcome. Participants that did not undergo two transseptal punctures were not included in this analysis.
Time Frame: 0-60 minutes (summation of first transseptal and second transseptal times)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Baylis RF Needle | Baylis Versacross RF Wire
Number analyzed (Participants) | 30 | 35
minutes | 20.5 [14 to 27.7] | 14.0 [10.6 to 15.6]

4. Secondary Outcome: Fluoroscopy Time
Description: Fluoroscopy time (amount of time operators used fluoroscopy during a transseptal puncture) was recorded for each participant, starting with insertion of the long guidewire into the femoral short sheath (J wire for RF needle group, VersaCross wire for RF wire group) and stopping once the transseptal sheath was positioned in the LA and the dilator and guidewire were fully removed from the long sheath. Median fluoroscopy time during the first and second transseptal punctures between the RF needle and RF Wire group was compared as a secondary outcome.
Time Frame: 0-60 minutes (from insertion of guidewire to removal of guidewire of first transseptal and second transseptal)
Population: All participants randomized underwent a first transseptal puncture. 6 patients from the RF needle group and 4 patients in the RF wire group did not undergo a 2nd transseptal puncture.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Baylis RF Needle | Baylis Versacross RF Wire
Number analyzed (Participants) | 36 | 39
minutes
  1st Transseptal | 2.0 [1.6 to 3.2] | 1.8 [1.3 to 2.2]
  2nd Transseptal: number analyzed (Participants) | 30 | 35
  2nd Transseptal | 2.4 [1.6 to 3.5] | 1.8 [1.5 to 2.7]

5. Secondary Outcome: Number of Participants With Equipment Exchanges
Description: An equipment exchange was defined as the removal of the J or RF wire from the dilator and sheath assembly before transseptal puncture; all RF needle punctures required at least 1 equipment exchange, although further exchanges could be performed as necessary if the initial pull-down resulted in inadequate positioning of the sheath and dilator and readvancement of the transseptal assembly into the SVC was necessary.
  The number of equipment exchanges during the cardiac ablation procedure between the RF need and RF wire groups were compared.
Time Frame: (0-8 hours) duration of cardiac ablation procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Baylis RF Needle | Baylis Versacross RF Wire
Number analyzed (Participants) | 36 | 39
Participants
  Number of exchanges = 0 | 0 | 37
  Number of exchanges = 1 | 26 | 0
  Number of exchanges = 2 | 5 | 2
  Number of exchanges >= 3 | 5 | 0

6. Secondary Outcome: Complication Rates
Description: The number of participants with complications during the procedure between the RF needle and RF wire groups was compared as a secondary outcome.
Time Frame: complications were assessed during the duration of cardiac ablation procedure (up to 8 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Baylis RF Needle | Baylis Versacross RF Wire
Number analyzed (Participants) | 36 | 39
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 1 year
Arm/Group | Baylis RF Needle | Baylis Versacross RF Wire
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/39
Other Adverse Events (participants affected / at risk) | 1/36 | 0/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baylis RF Needle (N=36) | Baylis Versacross RF Wire (N=39)
Procedure Complications (temporary AV Block) (Cardiac disorders) | 1 (1) | 0 (0) — 1 participant in the needle group had a mechanical injury to the atrioventricular (AV) node and transient ventricular asystole due to AV block, requiring brief pacing, resolved during procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT04645342/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT04645342/ICF_001.pdf